CLINICAL TRIAL: NCT02138903
Title: A Cardiac Ultrasound Evaluation of Two Types of Weaning Trials of Mechanical Ventilation for a First Weaning Trial
Acronym: CARWEAN
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-189; 2013-000960-26
Record Dates: First submitted 2014-04-11; First posted 2014-05-15 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Critical Care; Weaning of Mechanical Ventilation; Trans-thoracic Echocardiography; Mitral Doppler; Diastolic Function
Keywords: weaning; Cardiac; Echocardiography; Mechanical Ventilation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- ZEEP and tubing-spontaneous ventilation: Prospective clinical study in ICU with ventilated patients eligible to weaning trials of mechanical ventilation (ZEEP and tubing-spontaneous ventilation) comparing hemodynamic and cardiac effects evaluated by trans-thoracic echocardiography.
  Interventions: Other: trans thoracic echocardiography
- trans-thoracic echocardiography: Prospective clinical study in ICU with ventilated patients eligible to weaning trials of mechanical ventilation (ZEEP and tubing-spontaneous ventilation) comparing hemodynamic and cardiac effects evaluated by trans-thoracic echocardiography.
  Interventions: Other: trans thoracic echocardiography

INTERVENTIONS:
Other: trans thoracic echocardiography

SUMMARY:
Comparing the hemodynamic and cardiac effects of two types of weaning trials of mechanical ventilation in ICU patients of two French ICU.

DETAILED DESCRIPTION:
Prospective clinical study in ICU with ventilated patients eligible to weaning trials of mechanical ventilation (ZEEP and tubing-spontaneous ventilation) comparing hemodynamic and cardiac effects evaluated by trans-thoracic echocardiography.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ventilated requiring first weaning trial of mechanical ventilation

  * Stable respiratory and hemodynamic conditions
  * Consent of patients or family
  * Arterial line
  * Ventilated patients

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patients
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2014-01; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
left ventricular filling pressure | after 1 hour
  Echo-cardiographic evaluation is realized at the end of the weaning trial (1 hour) or less if failed

SECONDARY OUTCOMES:
Comparison of other echocardiographic parameters of left ventricular filling pressures | after 1 hour
  Comparison of other echocardiographic parameters of left ventricular filling pressures (E, Ea, deceleration time) at the end of weaning trial

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien PERBET, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France